CLINICAL TRIAL: NCT03750669
Title: Sequential Use of Nab-paclitaxel Plus Gemcitabine and mFOLFIRINOX as Neoadjuvant Chemotherapy for Resectable Pancreatic Cancer: A Randomized Control Study
Brief Title: Sequential Use of AG and mFOLFIRINOX as Neoadjuvant Chemotherapy for Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Liang Tingbo, Director of HBP Surgery, The Second Affiliated Hospital Zhejiang University School of Medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISPD-1
Record Dates: First submitted 2018-11-17; First posted 2018-11-23 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma Resectable; Neoadjuvant Chemotherapy
Keywords: Pancreatic Cancer; Pancreatic Adenocarcinoma; Gemcitabine; Nab-paclitaxel; Modified Folfirinox; Sequential treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Folic Acid; Fluorouracil; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant Chemotherapy (Experimental): Patients receive the sequential neoadjuvant chemotherapy of AG regimen (nab-paclitaxel plus gemcitabine) and mFOLFIRINOX before resection.
  Interventions: Drug: AG regimen; Drug: mFolfirinox
- control (No Intervention): Patients receive surgical treatment without any neoadjuvant treatments.

INTERVENTIONS:
Drug: AG regimen — Combination of Nab-paclitaxel 125 mg/m^2 and Gemcitabine 1000 mg/m^2
  Other Names: Nab-paclitaxel and Gemcitabine
  Arms: Neoadjuvant Chemotherapy
Drug: mFolfirinox — Folic acid 400mg/m^2, 5- fluorouracil 2400mg/m^2 for 46h, irinotecan 135mg/m^2 and oxaliplatin 68mg/m^2
  Other Names: Folic acid, 5- fluorouracil, irinotecan and oxaliplatin
  Arms: Neoadjuvant Chemotherapy

SUMMARY:
The prognosis of pancreatic cancer is extremely poor. Current guidelines recommend Nab-paclitaxel, Gemcitabine and modified Folfirinox as the first-line chemotherapeutic regimen. Studies have shown that sequential chemotherapeutic regimen can effectively delay the drug resistance and improve the effect of chemotherapy. Here investigators intend to assess the effect of sequential treatment with Nab-paclitaxel plus Gemcitabine and modified Folfirinox as neoadjuvant chemotherapy for resectable pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Investigators chose resectable pancreatic adenocarcinoma patients. The planned treatment was given to the participants after randomization. Tumor size, event-free survival, overall survival, drugs related side effects and other endpoints events were recorded and analyzed, to assess the sequential treatment with Nab-paclitaxel plus Gemcitabine and modified Folfirinox could or couldn't benefit the prognosis of resectable pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed pancreatic ductal adenocarcinoma (PDAC).
* No evidence of distant metastasis (such as liver, peritoneum, lung) evaluated by abdominal contrast-enhanced CT, MRI, and chest CT. PET/CT or other imaging examinations would be used if necessary.
* Initial assessment for definitive resectable tumors (resectability judgment is based on CT enhanced scan or magnetic resonance imaging, NCCN2018 first edition standard).
* ECOG score 0 or 1.
* Serum creatinine level is normal, and serum total bilirubin level is less than 1.5 x ULN.
* ALT and AST are less than 2 x ULN.
* If biliary obstruction is observed, biliary decompression should be performed when the patient is randomly assigned to receive neoadjuvant chemotherapy.
* Leukocyte count (> 3.5 x 10^6 /mL), neutrophil count (> 1.5 x 10^6 /mL), platelet count (> 80 x 10^6 /mL), hemoglobin (> 9 g/dL).
* Signed informed consent.

Exclusion Criteria:

* History of malignance treatment in the past, excluding basal and cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma
* Tumor is a local recurrent lesion.
* Imaging confirmed severe portal hypertension / cavernous transformation.
* Ascites
* Gastric outlet obstruction
* Respiratory failure requires supplementation of oxygen.
* Immune deficiency syndrome, such as active tuberculosis and HIV infection.
* Hematological precancerous diseases, such as myelodysplastic syndromes.
* Major cardiovascular diseases (including myocardial infarction, unstable angina, congestive heart failure, severe uncontrolled arrhythmia) during the past six months of enrollment.
* Evidence of clinical-related or previous interstitial lung disease, such as noninfectious pneumonia or pulmonary fibrosis, or baseline chest CT scan or chest X-ray findings
* Previous or physical findings of central nervous system disease, except for adequately treated (e.g. primary brain tumors, uncontrolled seizures or strokes with standard medications)
* Preexisting neuropathy > 1 (NCI CTCAE).
* Allograft requires immunosuppressive therapy or other major immunosuppressive therapies.
* Severe serious wounds, ulcers or fractures.
* Confirmed coagulant disease.
* Clinical evaluation is unacceptable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
event-free survival (EFS) | From randomization to any of the following events: progression of disease that precludes resection, local or distant recurrence, or death due to any cause, whichever occurs first. Up to approximately 60 months.
  Event-Free Survival assessed by the investigator according to RECIST 1.1 by investigator, defined as the time from randomization to any of the following events: progression of disease that precludes resection, local or distant recurrence, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | From randomization to death due to any cause. Up to approximately 60 months.
  Overall survival, the time from randomization to death due to any cause
Objective response rate | From randomization to the end of neoadjuvant therapy. Up to approximately 60 months.
  The proportion of patients with tumor size reduction of a predefined amount and for a minimum time period
Carbohydrate antigen 19-9 | Up to approximately 60 months
  Serum Carbohydrate antigen 19-9 level
Serious adverse events incidence | Up to approximately 60 months
  The proportion of patients with grade 3/4 adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, MD PhD, Principal Investigator — Department of HBP Surgery, SAHZJU
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided